CLINICAL TRIAL: NCT06475118
Title: Comparison of Serum Myokine Dosages and Imaging Methods in the Evaluation of Sarcopenia in Patients With Hepatocellular Carcinoma
Acronym: Myomachia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PA24055
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Sarcopenia; Hepatocellular Carcinoma
Keywords: Sarcopenia; Hepatocellular Carcinoma; myokines
MeSH Terms: conditions — Sarcopenia; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with hepatocellular carcinoma (Experimental)
  Interventions: Other: Dynamometry measurement, myokine dosing, sarcopenia calculation

INTERVENTIONS:
Other: Dynamometry measurement, myokine dosing, sarcopenia calculation — Blood sampling during standard pre-therapeutic care (at the same time with a standard blood testing) and dynamometry measurement. Retrieval of scanographic imaging and calculation of the L3 SMI index

SUMMARY:
It is known that some substances present in the blood, called 'myokines,' influence muscle loss. Some may accelerate this loss, while others may prevent it. Inflammatory substances in the blood can also contribute to muscle loss. Sarcopenia is assessed by an imaging technique called 'Skeletal Muscle Mass Index (SMI)' to measure muscle mass. This analysis can be done from radiological examinations. Sarcopenia has a serious impact on patients with hepatocellular carcinoma. It increases the risk of death, cancer recurrence, and decreases the response to treatments. Therefore, the investigators want to determine if blood tests for myokines obtained by simple blood draw can improve the assessment of sarcopenia in this specific setting.

DETAILED DESCRIPTION:
Background:

Sarcopenia, which is a reduction of muscle mass and function, frequently occurs from the age of 40 and is exacerbated by diseases such as cirrhosis, chronic inflammation, and cancer. It is well established that sarcopenia impairs quality of life and promotes the occurrence of complications. Myostatin, a muscle hormone (myokine), contributes to sarcopenia by promoting muscle degradation. Conversely, follistatin, an antagonist of myostatin, may play a role in maintaining muscle mass and protein synthesis. Irisin, another myokine, can protect against muscle atrophy and improve metabolism. Inflammatory cytokines like TNF-α and IL-6 can also contribute to sarcopenia by promoting muscle degradation. To evaluate sarcopenia in patients with cirrhosis and cancer, the most commonly used method is the calculation of the Skeletal Muscle Index (SMI) at the third lumbar vertebra (L3 SMI: Total Muscle Surface at L3 in cm²/ Height in m²). Other methods can also be used, but are susceptible to being influenced by water retention, particularly in cirrhotic patients. In patients with cirrhosis, sarcopenia negatively impacts quality of life and is associated with an increased risk of serious complications. In patients with hepatocellular carcinoma (HCC), it increases mortality, tumor recurrence, and reduces the response to treatments. Thus, its assessment and management are essential to improve the quality of life and prognosis of these patients. The validation of biological diagnostic criteria for sarcopenia would facilitate diagnosis and ensure follow-up without resorting to repetitive imaging.

Materials and Methods:

Type of study: Prospective validation study of a diagnostic method

Judgment criteria:

* Serum concentrations of myostatin, follistatin, and irisin
* Muscle surface calculated at L3 and parameterized according to height (L3 SMI)
* Muscle strength assessed by dynamometry

Investigation plan:

1. Screening of Patient after discussion in Multidisciplinary Liver Cancer Board
2. Proposal of the study during the announcement consultation after RCP.
3. Blood sampling during standard pre-therapeutic care and dynamometry measurement
4. Retrieval of scanographic imaging and calculation of the L3 SMI index
5. Blood dosages of myokines
6. Statistical analyses

Schedule:

* April 2024-July 2024: CPP evaluation
* August 2024-July 2025: Inclusion period.
* August 2024-July 2025: Radiological analyses (in parallel with the inclusions). Selection of available imagery, extraction of key images. Analysis of muscle mass and calculation of the L3 SMI index.
* August 2024-July 2025: Biological analyses (in parallel with the radiological analyses). Measurement of blood concentrations of myokines.
* August 2025-April 2026: Statistical analyses and article writing.

Expected Results and Prospects:

The current priority og investigators is to validate rapid and effective serum markers to facilitate the early diagnosis and clinical follow-up of sarcopenia in patients with hepatocellular carcinoma. In the long term, the goal is to implement early interventions aimed at mitigating the effects of sarcopenia. These serum markers could improve the management of liver diseases and cancers as key prognostic factors. The results of this study will also contribute to a better pathophysiological understanding of sarcopenia in these patients.

ELIGIBILITY:
Inclusion criteria:

* New diagnosis of HCC made by radiology and/or histopathology according to EASL criteria, regardless of the degree of hepatic fibrosis (METAVIR F0-F4)
* Availability of a pre-therapeutic three-phase contrast-enhanced abdominal-pelvic CT scan.

Non-inclusion criteria:

* Presence of an active cancer other than HCC
* Uncontrolled HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2025-11-22 (Estimated); Study Completion 2026-05-22 (Estimated)

PRIMARY OUTCOMES:
Determine if serum myokines measured in patients with HCC are correlated with muscle mass index assessed by standard scanographic technique. | Day 1
  Analysis of correlation between serum myokines measured in patients with HCC and muscle mass index assessed by standard scanographic technique

SECONDARY OUTCOMES:
Determine the serum myokine concentration threshold for the diagnosis of sarcopenia defined by an L3 SMI < 50 cm2/m2 in men | Day 1
  Analysis of correlation between serum myokines thresholds in patients with HCC and sarcopenia defined by an L3 SMI < 50 cm^2/m^2 in men
Determine the serum myokine concentration threshold for the diagnosis of sarcopenia defined by an L3 SMI < 39 cm2/m2 in women | Day 1
  Analysis of correlation between serum myokines thresholds in patients with HCC and sarcopenia defined by an L3 SMI < 39 cm^2/m^2 in women
Determine if serum myokines measured in patients with HCC are correlated with muscle strength assessed by dynamometry | Day 1
  Analysis of correlation between serum myokines measured in patients with HCC and Muscle strength assessed by dynamometry
Determine if inflammatory cytokines (IL6, TNFα) measured in patients with HCC are correlated with muscle mass index assessed by the standard scanographic technique | Day 1
  Analysis of correlation between inflammatory cytokines (IL6, TNFα) measured in patients with HCC and muscle mass index assessed by the standard scanographic technique

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France